CLINICAL TRIAL: NCT02040012
Title: A Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZP-531 in Healthy Volunteers, Overweight/Obese Volunteers and Patients With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate AZP531 in Healthy Volunteers, Overweight/Obese Volunteers and Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alizé Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AZP01-CLI-001
Record Dates: First submitted 2014-01-17; First posted 2014-01-20 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — cyclic des-acyl ghrelin (6-13)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZP-531 (Active Comparator): subcut administration once or twice daily
  Interventions: Drug: AZP-531
- Mannitol (Placebo Comparator): subcut administration once or twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZP-531
  Arms: AZP-531
Drug: Placebo
  Arms: Mannitol

SUMMARY:
Objectives:

Primary Objectives

* To investigate the safety and tolerability of single ascending doses of AZP- 531 in healthy volunteers.
* To investigate the safety and tolerability of single and multiple ascending doses of AZP-531 in overweight/obese volunteers.
* To investigate the safety and tolerability of single and multiple ascending doses of AZP-531 in patients with type 2 diabetes mellitus.

Secondary Objectives • To determine the plasma pharmacokinetic (PK) profile of AZP-531 after single and multiple doses.

Exploratory Objectives

• To obtain exploratory data on the effects of AZP-531 on the pharmacodynamic (PD) markers of blood glucose, interstitial glucose, insulin, and plasma acylated ghrelin (AG) and unacylated ghrelin (UAG)

ELIGIBILITY:
Inclusion Criteria:

* Part A: Healthy male volunteers, aged 18 to 50 years (inclusive) with a body mass index (BMI) of 20 to 28 kg/m2 (inclusive).
* Part B: Female (of non-childbearing potential) and male overweight/obese volunteers, aged 18 to 65 years (inclusive) with a BMI of 28 to 38 kg/m2 (inclusive).
* Part C: Female (of non-childbearing potential) and male patients with a confirmed diagnosis of type 2 diabetes mellitus for at least 3 months

Exclusion Criteria:

* Part A: Females and male volunteers who smoke and/or use other nicotine products within 6 months of screening are excluded.
* Part B: Current or ex-smokers with a smoking history of greater than 10 pack years (1 pack year = 20 cigarettes smoked per day for 1 year) and any clinically significant abnormalities in physical examination, electrocardiogram (ECG), clinical chemistry, haematology, coagulation or urinalysis results at screening or on admission, as judged by the Investigator.
* Part C: Current or ex-smokers with a smoking history of greater than 10 pack years (1 pack year = 20 cigarettes smoked per day for 1 year), any clinically significant abnormalities other than those attributed to type 2 diabetes mellitus in physical examination, ECG, clinical chemistry, haematology, coagulation or urinalysis results at screening or on admission, as judged by the Investigator, and estimated glomerular filtration rate <40 mL*min-1*1.73m-2 calculated by the Modification of Diet in Renal Disease formula.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
To investigate the number of adverse events of single and multiple ascending doses AZP-531 in healthy volunteers, in overweight/obese volunteers, in patients with type 2 diabetes mellitus. | 1 to 14 days

SECONDARY OUTCOMES:
To determine the plasma pharmacokinetic (PK) profile of AZP-531 after single and multiple doses | 1 to 14 days

OTHER OUTCOMES:
To obtain exploratory data on the effects of AZP-531 on the pharmacodynamic (PD) markers | 1 to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: James Ritter, MD Professor, Principal Investigator — Quintiles Drug Research Unit at Guy's Hospital
Locations (1):
- Quintiles Drug Research Unit at Guy's Hospital, London, London, United Kingdom